CLINICAL TRIAL: NCT01371019
Title: Proteomic Assessment of Preterm Birth
Acronym: PAPR
Status: Completed | Type: Observational
Sponsor: Sera Prognostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Sera - 004
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Preterm Birth
Keywords: Preterm Birth, Proteomics
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with preterm delivery
- Women without preterm delivery

SUMMARY:
The purpose of this study is to to collect and store blood samples that will be utilized to develop a multimarker test to predict preterm delivery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older.
* Subject has a singleton pregnancy.
* Subject is able to provide consent.

Exclusion Criteria:

* Subject is pregnant with more than one fetus.
* There is a known or suspected fetal anomaly.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who are receiving prenatal care.
Sampling Method: Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Spontaneous Preterm Birth | August 2015

CONTACTS AND LOCATIONS:
Overall Officials: Durlin E Hickok, MD, MPH, Study Director — Sera Prognostics, Inc.
Locations (13):
- United States (13):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - San Diego Perinatal Clinic, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - Baystate Medical Center, Springfield, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Intermountain Medical Center Suite 100, 5121 S. Cottonwood Street ,, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - LDS Hospital, Salt Lake City, Utah

REFERENCES:
- [Background] Esplin MS, Merrell K, Goldenberg R, Lai Y, Iams JD, Mercer B, Spong CY, Miodovnik M, Simhan HN, van Dorsten P, Dombrowski M; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Proteomic identification of serum peptides predicting subsequent spontaneous preterm birth. Am J Obstet Gynecol. 2011 May;204(5):391.e1-8. doi: 10.1016/j.ajog.2010.09.021. Epub 2010 Nov 11. PMID 21074133